CLINICAL TRIAL: NCT07069231
Title: Effect of Bio-activation on Epithelial and Connective Cell Adhesion to Titanium Abutments: Split Mouth Clinical Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universita degli Studi di Genova (Other)
Responsible Party: Principal Investigator, Paolo Pesce, Prof., Universita degli Studi di Genova
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Abutment adhesion
Record Dates: First submitted 2025-07-05; First posted 2025-07-16 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Missing Tooth/Teeth
MeSH Terms: conditions — Anodontia

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Machined Abutment - control (No Intervention): The control group received MUA without plasma treatment.
- Plasma abutment - test (Experimental): .The MUA allocated to the test group will be placed in a plasma reactor (Plasmapp, South Korea) for decontamination and activation of the surface. In order to restrict any post-treatment contamination; abutments will be inserted immediately after the end of the plasma process.
  Interventions: Device: the test group were placed in an Argon plasma reactor

INTERVENTIONS:
Device: the test group were placed in an Argon plasma reactor — the test group were placed in an Argon plasma reactor
  Arms: Plasma abutment - test

SUMMARY:
The aim of this "in vivo" controlled trial is to assess soft tissue cell adhesion to titanium abutments subjected to different cleaning procedures - no treatment (as they come from the industry), and cleaning by plasma- at an early healing time.

In fact, the primary aim is Quantity and Quality of soft tissue adhesion at the microscopic level (e.g Fibronectin, Integrin-actin).

The secondary Aim - Clinical parameters and outcomes - BOP, PPD, MBL (Marginal Bone Level to check influence of plasmapp-treated abutments).

The null hypothesis of the study was that the cleaning procedure applied to implant abutments has no effect on soft tissue cell adhesion and MBL at an early healing time.

ELIGIBILITY:
Inclusion Criteria:

* presence of at least 4 mm of keratinized mucosa around the implants,
* patients aged 18 years or older
* medically healthy patients (ASA I), or patients with mild systemic disease (ASA II)
* Total or partial edentulous state with space for at least 2 implants

Exclusion Criteria:

* ASA physical status 3
* severe smokers (> 10 cig/day)
* patients undergoing bisphosphonate therapy
* pregnant or lactating women
* estrogen-related hormonal disorders or hormonal substitution therapy patients with a history of head and neck cancers and radiotherapy in this region

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-07-15 (Estimated); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
connective tissue coverage | 3 months post-op
  • Coverage was defined as the extent to which the abutment surface was occupied by adherent cells. It reflects the spatial distribution of cells across the surface, providing a measure of surface colonization.
  Coverage was independently scored on a scale from 1 to 10 by two blinded operators who were unaware of the sample group assignments (i.e., activated vs control). The individual scores were subsequently averaged to obtain a representative value for each parameter per sample.

SECONDARY OUTCOMES:
Connective tissue density | 3 months post-op
  • Density was defined as the degree of cellular accumulation in the regions where cells were present. This parameter reflects the local compactness of cells, irrespective of how widely they are spread across the surface.
  Density was independently scored on a scale from 1 to 10 by two blinded operators who were unaware of the sample group assignments (i.e., activated vs control). The individual scores were subsequently averaged to obtain a representative value for each parameter per sample.
Mean bon loss | 1 year post-op
  MBL will be measured at 1-year follow up using orthopanoramic or endo-oral Xray.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Canullo L, Donato A, Savadori P, Radovanovic S, Iacono R, Rakic M. Effect of argon plasma abutment activation on soft tissue healing: RCT with histological assessment. Clin Implant Dent Relat Res. 2024 Feb;26(1):226-236. doi: 10.1111/cid.13286. Epub 2023 Oct 18. PMID 37853303